CLINICAL TRIAL: NCT00839735
Title: Trefoil Peptides in Lung Diseases
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Thomas Lund, MD, Bispebjerg Hospital
Other Study IDs: H-B-2008-120
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- COPD: Chronic obstructive pulmonary disease
- Asthma
- Healthy controls

SUMMARY:
The study focuses on trefoil family factor (TFF) peptides in sputum in lung diseases. The investigators hypothesize that TFF peptides are upregulated in lung diseases characterized by mucus hypersecretion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Informed consent

Exclusion Criteria:

* Upper and lower airway infection 2 weeks prior to visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic obstruction pulmonary disease (COPD) Subjects with asthma Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
TFF in sputum | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Lund, MD PhD, Principal Investigator — Respiratory and Allergy Research Unit
Locations (1):
- Respiratory and Allergy Research Unit, Department of Respiratory Medicine L, Bispebjerg Hospital, Copenhagen, Denmark